CLINICAL TRIAL: NCT05834855
Title: Non-inferiority Study of Rituximab Compared to Ocrelizumab in Relapsing Multiple Sclerosis
Brief Title: Non-inferiority Study of Rituximab Compared to Ocrelizumab in Relapsing MS
Acronym: Noisy Rebels
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Stichting Treatmeds (Unknown)
Responsible Party: Principal Investigator, Eva M.M. Strijbis, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Anti-CD20 in RMS
Record Dates: First submitted 2023-04-03; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Demyelinating Diseases
Keywords: ocrelizumab; rituximab; non-inferiority
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Demyelinating Diseases | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled double-blind non-inferiority trial in The Netherlands
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient, site personnel administrating infusions, and the treating and evaluating neurologist and study nurse will all be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ocrelizumab (No Intervention): The standard group will receive ocrelizumab (600 mg, the first dosage given in two infusion of 300 mg with a two week interval) following the current treatment protocol
- Rituximab (Experimental): The experimental group will receive rituximab (1000 mg). Rituximab will be given intravenously. To ensure blinding of treatment allocation two dosages of 500 mg with a two week interval will be given instead of one initial dosage of 1000 mg of rituximab to mimic the ocrelizumab protocol
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Treatment with rituximab
  Other Names: MabThera; Truxima; Ruxience; Rixathon
  Arms: Rituximab

SUMMARY:
Rationale: Ocrelizumab is widely and effectively used to treat relapsing multiple sclerosis (RMS). Phase II studies and data from large patient cohorts indicate that rituximab, another anti-CD20 monoclonal antibody, is probably equally effective and safe as ocrelizumab in the treatment of RMS. An advantage of rituximab is a considerably lower price. Therefore we will start a study aimed at demonstrating non-inferiority of rituximab compared to ocrelizumab in RMS. If non-inferiority of rituximab can be shown, important reductions in the cost of treatment of RMS will be possible, without loss of efficacy.

Objective: Evaluating the efficacy and safety of ritixumab compared to ocrelizumab in the treatmens of RMS.

Study design: Randomized double blind multi-centre non-inferiority study of rituximab compared to ocrelizumab in 200 patients with RMS. The trial duration will be 30 months

Study population: The study population consists of 200 adult RMS patiens with an indication to start anti-CD20 monoclonal antibody treatment.

Intervention: Patients will be randomized 1:1 into the standard group (ocrelizumab treatment) or the experimental group (rituximab treatment).

Main study parameters: To conclude non-inferiority of rituximab there will be one primary endpoint: the proportion of patients free of inflammatory disease activity (defined as: new or enlarged T2 lesions) between week 24 (M6) and week 96 (M24) of treatment in each arm. Secondary trial endpoints are presence and number of clinical relapses,T2 and contrast enhancing lesion volumes, brain volume and brain volume changes, disease progression (defined as clinically relevant change on any of the measures: EDSS, T25FW, 9HPT, SDMT), biochemical parameters such as lipidomics and neurofilament light (NfL), immunological parameters, safety as measured by the number of (serious) adverse events ((S)AE), quality of life (EQ-5D-L) and treatment satisfaction (TSQM) and patient reported measures of MS impact (MSIS-29) and well-being (questionnaire on physical complaints)

Nature and extent of the burden and risk: Patients included in this study will be treated and monitored by MRI, clinical tests and laboratory tests according to existing protocols and will not be exposed to extra or unknown risks. They will have extra annual questionnaires and larger blood samples at some time points. There is extensive experience with both rituximab and ocrelizumab as efficacious and safe treatments of RMS.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 years and older
2. A diagnosis of relapsing MS according to the 2017 revised diagnostic criteria
3. Indication to start treatment with anti-CD20 therapy according to the treating neurologist and the relevant label in the Netherlands for treatment of relapsing MS
4. Able to understand written and spoken Dutch or English
5. Capable of giving signed informed consent including compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
6. Screening EDSS score ≤ 6.5 .

Exclusion Criteria:

Medical Conditions

1. A known allergy or other intolerability to RTX, OCR, gadolinium-based MRI contrast agents, or corticosteroids.
2. A diagnosis of primary progressive MS according to the diagnostic criteria.
3. A diagnosis of not-active secondary progressive MS.
4. Chronic infectious diseases such as tuberculosis, VZV, hepatitis virus or HIV, as well as hepatitis B surface antigen positivity and/or hepatitis C PCR positivity verified at screening visit.
5. A history of proven inflammatory bowel disease such as M. Crohn or ulcerative colitis
6. Prior or current psychiatric illness, mental deficiency or cognitive dysfunction influencing the patient ability to make an informed consent or comply with the treatment and follow-up phases of this protocol.
7. Cardiac disease that makes treatment with OCR or RTX contra-indicated as stated by the most recent SmPC
8. Active malignancy or prior history of malignancy that makes treatment with OCR or RTX contra-indicated as stated by the most recent SmPC.
9. WBC < 1.5 x 109/L if not caused by a reversible effect of documented ongoing medication. If caused by a reversible effect of documented ongoing medication the WBC count must be > 1,5 x 109/L before start of study treatment.
10. Platelet (thrombocyte) count < 100 x 109/L
11. ALAT and/or ASAT more than 2 times the upper normal reference limit (ULN)
12. Serum creatinine > 200 μmol/L
13. Serum bilirubin > ULN
14. Serum IgG < LLN
15. Pregnant or breast-feeding women
16. Women of childbearing potential (WOCBP) not able or willing to use highly effective methods of birth control per ICH M3 (R2) that result in failure rate of ≤ 1% per year when used consistently and correctly for the duration of the study OR until 3 months after last dose administered.
17. History of serious or life-threatening infusion reaction to OCR or RTX
18. Treatment with glucocorticoids or ACTH within one month prior to start of study treatment

    Prior/Concomitant Therapy
19. Previous use of second line MS-therapies cladribine, RTX, alemtuzumab, OCR, ofatumumab, hematopoietic stem cell therapy (HSCT) or other immunosuppression therapies with long lasting effects. Mitoxantrone is allowed if used > 1 year before enrolment. If any of these medications have been used for indications other than MS, patients can be included if the medications have not been used the year before enrolment. Previous treatment with natalizumab is allowed if the reason to switch was disease activity (so not allowed in for example cases that switch from natalizumab to anti-CD20 therapy because of JCV positivity).
20. Concomitant use of systemic immunosuppressive medication (except corticosteroids for symptomatic treatment of relapses).

    Prior/Concurrent Clinical Study Experience
21. Currently enrolled in another investigational device or drug study, or less than 30 days since ending of another investigational device or drug study (s), or receiving other investigational treatment(s). Patients participating in a purely observational studies will be allowed to participate.

    Lifestyle
22. Current alcohol or drug dependencies.

    Diagnostic assessments
23. Presence of metallic objects implanted in the body, that would preclude the ability of the patient to safely have MRI exams.
24. Not willing to undergo MRI scans with i.v. gadolinium injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients free of inflammatory disease activity | between month 6 and month 24
  Proportion of patients with no new or enlarged T2 lesions on brain MRI between month 6 and month 24

SECONDARY OUTCOMES:
Presence and number of clinical relapses | Baseline, month 6, month 24
  Clinical relapses during treatment
Contrast enhancing lesions | Baseline, month 6, month 24
  Proportion of patients with no contrast enhancing lesions on brain MRI
Average number of T2 lesions on brain MRI | Baseline, month 6, month 24
  The average number of new/enlarged T2 lesions between baseline, month 6 and month 24 on brain MRI
Disability progression during follow-up | Baseline, month 6, month 24
  Disability progression measured on the Expanded Disability Status Scale (EDSS)
Disability progression during follow-up | Baseline, month 6, month 24
  Disability progression measured on the timed 25 foot walk test (T25FW)
Disability progression during follow-up | Baseline, month 6, month 24
  Disability progression measured on the Nine Hole Peg Test (9HPT)
Disability progression during follow-up | Baseline, month 6, month 24
  Disability progression measured on the Symbol Digit Modalities Test(SDMT)

OTHER OUTCOMES:
Anti-drug antibodies | 30 months
  Proportion of patients with anti-drug-antibodies during 30 months of treatment
Infusion reactions | 30 months
  Proportion of patients with immediate and delayed infusion reactions during 30 months of treatment
Infections | 30 months
  Proportion of patients with infections during 30 months of treatment
Malignancies | 30 months
  Proportion of patients with malignancies during 30 months of treatment
Adverse events | 30 months
  Proportion of patients with any SAE/SAR and AESI during 30 months of treatment
Burden of physical senstations during treatment | Baseline, month 6, month 12, month 18, month 24, month 30
  Burden of physical sensations prior to, after, and between infusions as measured with wearing-off questionnaire and question 5 of the RAPID3-HAQ2 questionnaire
Quality of life questionnaires | Baseline, month 6, month 12, month 18, month 24, month 30
  Quality of life as measured by multiple sclerosis impact scale-29 (MSIS-29)
Quality of life questionnaires | Baseline, month 6, month 12, month 18, month 24, month 30
  Quality of life as measured by EuroQol-5 Dimension (EQ-5D)
Treatment satisfaction | Baseline, month 6, month 12, month 18, month 24, month 30
  Treatment satisfaction as measured with the Treatment Satisfaction Questionnaire Measurement (TSQM)
Lymphocytes | 30 months
  Absolute numbers of different lymphocyte subsets prior to infusion during 30 months of treatment
Neurofilament | 30 months
  Serum levels of neurofilament during 30 months of treatment
Dynamics of B-cell depletion | Baseline, week 2, month 6, month 12, month 18, month 24, month 30
  B-cell count (thousand/ml) (normal range: 100-300 thousand/ml)
Dynamics of B-cell repopulation | Baseline, week 2, month 6, month 12, month 18, month 24, month 30
  B-cell count (thousand/ml) (normal range: 100-300 thousand/ml)
Dynamics of ocrelizumab drug concentrations | Baseline, week 2, month 6, month 12, month 18, month 24, month 30
  Dynamics of ocrelizumab drug concentrations (microgram/mL)
Immunoglobulins | Baseline, week 2, month 6, month 12, month 18, month 24, month 30
  Serum levels of immunoglobulins
Serum levels | 30 months
  Serum levels of chemokines and cytokines, protectins, resolvins, maresins, and lipoxins during 30 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bob van Oosten, Dr, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, location VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After medical ethical commitee approved the study protocol